CLINICAL TRIAL: NCT00934349
Title: Determination Study of Dry Beriberi in Patients Native to the Comoro Archipelago, in Mayotte (MABECO).
Brief Title: Study of Dry Beriberi in Mayotte, Comoro Archipelago
Acronym: MABECO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Groupe Hospitalier Sud Reunion (Other)
Responsible Party: Joaquin MARTINEZ / Clinical Research and Innovation Director, Regional Hospital, Reunion Island
Other Study IDs: 2009-A00348-49; CHR-GHSR_2009-03/01
Record Dates: First submitted 2009-07-02; First posted 2009-07-08 (Estimated); Last update posted 2009-07-08 (Estimated); Status verified 2009-07

CONDITIONS: Dry Beriberi
Keywords: Comoro Island; vit B1 intake; Thiamine status; Genetic factor

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples drawn for thiamine status, vit B1 dosage will be centrifuged and a serum sample will be frozen at -20°C, transferred to Regional Hospital of Reunion Island - GHSR and retained in virology laboratory of Dr MICHAULT after end of study for further explorations on beriberi
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Patient: Native to the Comoro Archipelago (Grande Comore, Mayotte, Anjouan, Mohéli) fulfilling the clinical definition of the dry beriberi.
- Control: Native to the Comoro Archipelago, living in the same household as the patient, sharing the same meals. Free from beriberi and with normal neurological examination.

SUMMARY:
The purpose of this study is to assess the existence of a genetic factor, suspected to be involved, aside from likely food deficiency contribution, in occurrence of dry beriberi, in patients who experienced dry beriberi and in a case group composed of 3 people, free from beriberi, within the same household.

DETAILED DESCRIPTION:
A team of 2 investigators, a nurse and an investigator speaking French, Shibushi and Shimaore (3 languages in use in Mayotte), will visit exposed patients who agreed to participate to the study.

3 controls, fulfilling inclusion criteria, will be recruited within the household by drawing lots.

Clinical examination and food survey by means of a questionnaire will be performed.

Blood samples will be drawn to determine thiamine status, vitamin B1 dosage, erythrocyte transketolase activity and thiamine pyrophosphate effect, analysis will be performed by Biomnis laboratory in Lyon.

For the genetic study, 4 drops of blood will be put down on Whatman paper and sent to Dr Johannes COY in Darmstadt Germany, for DNA extraction and PCR screening for mutations.

ELIGIBILITY:
Inclusion Criteria:

* patients
* Native to the Comoro Archipelago (Grande Comore, Mayotte, Anjouan, Mohéli)
* Fulfilling the clinical definition of the dry beriberi.
* Both sexes.
* Older than 15 years and 3 months (limit of the paediatrics).
* Having signed and whose legal representatives signed the form of assent, having understood the information.
* Benefiting from a social coverage regime.
* Controls
* Native to the Comoro Archipelago.
* People living in the same household as the patient, sharing the same meals.
* Both sexes.
* Older than 15 years old and 3 months.
* Free from beriberi.
* With normal neurological examination.
* Having signed and whose legal representatives signed the form of assent, having understood the information.
* Benefiting from a social coverage regime.

Exclusion Criteria:

* Aged under 15-year-old and 3 months.
* For the patients and the witnesses, the presence of pathologies known to increase needs in vitamin B1 (cancer, infectious diseases, fever, hyperthyroïdism, chronic alcoholism).

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients Native to the Comoro Archipelago (Grande Comore, Mayotte, Anjouan, Mohéli) fulfilling the clinical definition of the dry beriberi. 3 controls fullfilling inclusion criteria will be recruited within the houshold by drawing lots.among
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2009-06

PRIMARY OUTCOMES:
Mutations on one of the alleles of the promoter of the gene TKTL1 (transketolase-like gene) in the homozygous state in the patients and not in the controls (heterozygotes or not carrier of the mutation). | day 1

SECONDARY OUTCOMES:
To evaluate food intakes in vitamin B1 and anti-thiamine factors (polyphenols). | day 1
To evaluate Thiamine biological status (blood thiamine, erythrocyte transketolase activity and the thiamine pyrophosphate effect) | day 1

CONTACTS AND LOCATIONS:
Overall Officials: ERIC DOUSSIET, PHD, Principal Investigator — Regional Hospital La Reunion - CIC-EC; IAN PERINET, PHD, Principal Investigator — CENTRAL HOSPITAL MAYOTTE; JULIETTE WOESSNER, PHD, Principal Investigator — CENTRAL HOSPITAL MAYOTTE; Francoise DARCEL, PHD, Study Director — Regional Hospital La Reunion - GHSR
Locations (1):
- Central Hospital - MAYOTTE, Mamudzu, France